CLINICAL TRIAL: NCT00416754
Title: Improving the Long-Term Outcomes of BRCA1/BRCA2 Mutation Testing
Brief Title: Genetic Counseling in Women at Risk for BRCA1 or BRCA2 Mutations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: CDR0000450754; R01CA082346 (NIH); P30CA051008 (NIH); GUMC-2000-305
Record Dates: First submitted 2006-12-27; First posted 2006-12-28 (Estimated); Last update posted 2017-04-07 (Actual); Status verified 2017-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; stage I breast cancer; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: counseling intervention — subjects will receive genetic counseling

SUMMARY:
RATIONALE: Genetic counseling and using an interactive computer program may help women at risk for breast cancer make medical decisions about treatment.

PURPOSE: This randomized clinical trial is studying standard genetic counseling to see how well it works when given together with or without a medical decision-making computer program in women at risk for BRCA1 or BRCA2 mutations.

DETAILED DESCRIPTION:
OBJECTIVES:

* Evaluate the impact of BRCA1/BRCA2 testing among members of hereditary breast-ovarian cancer families.
* Evaluate the long-term impact of genetic counseling and testing on psychosocial and behavioral outcomes.
* Evaluate the relative impact of standard genetic counseling (SGC) versus SGC plus the interactive decision-aid (IDA) on medical decision-making.
* Evaluate the relative impact of SGC vs SGC + IDA on psychological well-being.
* Explore the mechanisms by which the SGC + IDA intervention impacts on psychosocial and behavioral outcomes.

OUTLINE: This is a multicenter study.

Eligible women are asked to participate in a baseline telephone interview over 30 minutes and then invited to a genetic counseling session over 1.5-2 hours that includes information about BRCA1/2 testing. Patients are then offered BRCA1/2 testing, and the test results (i.e., mutation carrier vs noncarrier) are presented at a subsequent in-person individual genetic counseling session over 1.5-2 hours. Patients who tested positive for BRCA1 or 2 mutation are randomized to 1 of 2 counseling arms. All other patients proceed to follow up.

* Arm I (standard genetic counseling): No further counselor-initiated contact is scheduled.
* Arm II (individualized decision aid): Patients are asked to view an interactive computer program that is designed to help the patients make medical decisions based on their breast cancer risk.

Outcome assessments, including quality of life assessment, are conducted at 2, 6, and 12 months.

PROJECTED ACCRUAL: A total of 950 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Members of hereditary breast/ovarian cancer families (in which there is at least a 10-20% prior probability of a BRCA1/2 mutation) OR who have a first-degree relative with a known BRCA1 or BRCA2 mutation
* Prior diagnosis of breast cancer allowed

  * Must not be undergoing active treatment
  * Patients with prior bilateral mastectomy are eligible for study but not eligible for randomization

PATIENT CHARACTERISTICS:

* Female only
* No psychiatric or cognitive disorder that would preclude giving informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Ages: 25 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1109 (Actual)
Dates: Start 2000-12; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
patient satisfaction | 1 year
  subjects will complete questionnaires re; genetic counseling experience

CONTACTS AND LOCATIONS:
Overall Officials: Marc Schwartz, PhD, Principal Investigator — Lombardi Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No